CLINICAL TRIAL: NCT04020471
Title: How Variations in Patient Pharmacogenomic Profiles Affect Pain and Narcotic Requirements Following Total Knee Arthroplasty (TKA)
Brief Title: How Variations in Pharmacogenomic Profiles Affect Pain and Narcotic Needs Following Total Knee Arthroplasty (TKA)
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Richard Wixson, Physician, FPA, Endeavor Health
Other Study IDs: EH19-023
Record Dates: First submitted 2019-03-29; First posted 2019-07-16 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty (TKA)
Keywords: Pharmacogenomic Profile; Knee Osteoarthritis; Total Knee Arthroplasty (TKA); Narcotic Use
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: All subjects who have completed their standard of care total knee arthroplasty will undergo pharmacogenomics testing and will complete a daily pain and medication diary for 30 days post discharge from the hospital. Subjects will be offered a consultation visit with a member of the Pharmacogenomics Team to discuss results.
  Interventions: Other: Pain Scale/Medication Log

INTERVENTIONS:
Other: Pain Scale/Medication Log — Daily recording of pain level after surgery and recording of medication taken for pain relief.

SUMMARY:
The purpose of the study is to gain a better understanding of how genetic variations can affect pain experience and the need and type of pain control medication after a total knee replacement.

DETAILED DESCRIPTION:
The purpose of the study is to gain a better understanding of how genetic variations can affect pain experience and the need and type of pain control medication after a total knee replacement. People experience pain differently. The type and amount of medication required to control pain varies. Post-operative pain often requires narcotics to keep patients comfortable. It has been shown that there is a genetic difference in how people respond to pain and how they respond to the medications used for the relief of pain. Opioids are often used to relieve pain after surgery. These medications can be abused and have had a role in the current opioid crisis.

Pharmacogenomics is the study of how patients respond to and metabolize drugs and medications based on their genetic profiles. This study will collect data on the pain experienced by participants and the narcotics used after total knee replacements. This will be correlated with the participants' pharmacogenomic profiles obtained though DNA testing. There are no treatment interventions in this study. Although a pharmacogenomic profile will be obtained at the first post-operative visit and reported approximately 3 weeks later, the subject will have completed the need for pain relief. The study is expected to last 2 years with 300 subjects enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Unilateral primary Total Knee Arthroscopy (TKA)
* Knee Osteoarthritis
* Planned discharge to home

Exclusion Criteria:

* Unicompartmental Total Knee Arthroscopy (TKA)
* Revision Total Knee Arthroscopy (TKA)
* Knee flexion contracture > 15°
* Axial deformity > 15°
* Previous or current chronic narcotic use for pain > 3 months
* Previous or current substance abuse
* Any chronic pain condition
* Any dementia or cognitive disorder
* Discharge to Skilled Nursing Facility
* Rheumatoid arthritis
* Potential difficulty completing daily pain scores and medication use
* Previous NorthShore genotyping
* Currently taking CYP2D6 inhibitors (list in appendix)
* Currently taking CYP2D6 inducers (list in appendix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis who are scheduled for a primary total knee replacement and excluding those with significant deformity, partial knee replacement, and revision surgery.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Determine how variation in a pharmacogenomics panel affects a patient's perception of pain. | 30 days
  The variation in genetics will be investigated using a standard 20 gene clinical pharmacogenomics panel. Three of these genes (CYP2D6, OPRM1, and COMT) have effects on opioid metabolism, opioid transport, pain perception, and opioid receptors. The results of the pharmacogenomics panel in relation to pain as assessed by the VAS (Visual Analog Scale) numeric pain scale completed by each subject for maximum pain experienced with activity, average pain, and lowest level of pain over the previous 24 hours. The VAS is a self-reported score which measures pain on a 0-10 scale with 10 being the most amount of pain possible and 0 being no pain.
Determine how variation in a pharmacogenomics panel affects the amount of opioids needed to control a patient's pain. | 30 days
  The results of the pharmacogenomics panel in relation to the amount of opioids needed to control post-operative pain for the first month following surgery will be assessed via a daily medication log completed by patients where they record the specific medication and dose taken in the previous 24 hour period each day of the month following surgery. This will be converted to morphine milligram equivalents (MME) and expressed as the total MME used in the first post-operative month.

SECONDARY OUTCOMES:
A secondary outcome will be measuring changes in the KOOS Jr (Knee injury and Osteoarthritis Outcome Score- Junior). | 1 year
  Study subjects will complete the KOOS Jr questionnaire at pre-op, 4 months and 1 year after surgery. KOOS, Jr is scored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Secondary outcome will be measuring changes in ROM (range of motion) as determined by the physician. | 1 year
  The knee exam/ROM will be completed by the patient's surgeon at standard-of-care clinic visits pre-op, 1 month, 4 months, and 1 year after surgery.
Secondary outcome will be measuring changes in the PROMIS-43. | 1 year
  Subjects will complete the PROMIS-43 questionnaire at pre-op, 4 months and 1 year after surgery. The score comprises questions from seven domains: Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities as well as a numeric rating scale for pain from 0-10 with 10 being the worst. They may be reported as T-scores (difference compared to the population average, measure in standard deviations). A score of 50 is the average for the United States general population. For undesirable concepts such as Depression, a T-score of 60 is one standard deviation worse than average. Alternatively, a Depression T-score of 30 is two standard deviations better than average. For favorable concepts like Ability to Participate in Social Roles and Activities, a T-score of 60 is one standard deviation better than average while a T-score of 30 is two standard deviations worse than average.
Secondary outcome will be measuring changes in the VR-12 (Veterans Rand Item Health Survey). | 1 year
  Study subjects will complete the VR-12 at pre-op, 4 months and 1 year after surgery. The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The score encompasses questions from seven domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The interval score ranges from 0 to 100 where 0 represents mental or physical disability and 100 represents perfect mental or physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wixson, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided